CLINICAL TRIAL: NCT00683709
Title: Metabolic Side Effects, Diet and Exercise Counseling and Brain Function in a Naturalistic Clinical Trial of Clozapine for Treatment Resistant Bipolar and Schizoaffective Disorder
Brief Title: Specialized Clozapine Clinic for Bipolar and Schizoaffective Disorder
Status: Completed | Type: Observational
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Dr. Gary Hasey, McMaster University
Other Study IDs: 06-2726
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Bipolar Affective Disorder; Schizoaffective Disorder
Keywords: Bipolar and Schizoaffective Disorder; Clozapine; Metabolic Side Effects; Diet & Exercise; BMI
MeSH Terms: conditions — Bipolar Disorder; Psychotic Disorders; Motor Activity | interventions — Counseling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Counselling as Usual: Discussing Clozapine medication, diet and exercise as per clinical protocol potential weight changes
  Interventions: Behavioral: Counselling as Usual
- Cognitive Behavoural Therapy: Counselling about Clozapine medication, diet and exercise in a structured fashion using Cognitive Behavioural Therapy about potential weight changes
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: Counselling as Usual — 5 - 20 minutes, about the effects of clozapine on body weight, appetite, blood sugar and fats such as cholesterol and triglycerides in the blood, and how these might affect your health in the future.
  Groups: Counselling as Usual
Behavioral: CBT — 45 - 60 minutes individual treatment sessions focused on nutrition, exercise and weight control and will occur weekly for 4 weeks. After this, 10 group sessions focused on weight reduction will be held every 2 weeks. This will be followed by 6 group sessions focused on weight maintenance held every 2 weeks.
  Groups: Cognitive Behavoural Therapy

SUMMARY:
Bipolar Disorder (BD) and Schizoaffective Disorder (SA) clients.

* determine if after 12 months of treatment with clozapine, the BMI changes with clients who are councelled as usual regarding weight gain while on Clozapine.
* determine if after 12 months of treatment with clozapine, the BMI changes with intense, structured councelling about diet and exercise.

DETAILED DESCRIPTION:
To determine whether the changes in BMI produced in subjects with Bipolar Disorder (BD) and Schizoaffective Disorder (SA) by 12 months of treatment with clozapine, can be diminished after an intense and highly structured intervention focused on diet and exercise, compared with the usual brief counseling regarding weight gain on this drug.

ELIGIBILITY:
Inclusion Criteria:

* Clients diagnosed with bipolar disorder or schizoaffective disorder
* Clients who respond poorly to treatment
* Males and females ages 18 years or older
* Clients who have had a trial of antipsychotics, incl. at least one atypical antipsychotic plus at least 2 mood stabilizers
* Clients who are capable of providing informed consent

Exclusion Criteria:

* Clients who take carbamazepine
* Clients with a history of extremely low white blood counts
* Clients with severe kidney, liver or heart disease, or heart operation
* Clients are hypersensitive to clozapine
* Clients who have a history of serious side effects after previous treatment with clozapine
* Clients with alcohol or drugs abuse within the last 3 months
* Clients who have a seizure disorder
* Clients who have metal in the head, neck or eyes, shrapnel, bullets, or body piercing, a pacemaker, brain aneurism clips, cochlear implant, hearing aid, tens unit, spinal implant, or pregnancy. These safety measures are necessary because of the magnetic fields of the MRI scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric outpatients from within the catchment area of the hospitalwho suffer from chizoaffective disorder and respond poorly to treatment offered to participate in research
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2007-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Increases in BMI in subjects with BD and SA after 12 months of clozapine treatment will be smaller in subjects treated with CBT ex/diet compared with those receiving CAU. | 5 years

SECONDARY OUTCOMES:
Adverse changes in plasma lipids, blood sugar, and fitness level will be greater in subjects treated with CBT ex/diet compared with those receiving CAU after 12 months of clozapine treatment. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hasey, MD, Principal Investigator — St. Joseph's Healthcare and McMaster University, Hamilton
Locations (1):
- St. Joseph's Healthcare, Centre for Mountain Health Services, Hamilton, Ontario, Canada